CLINICAL TRIAL: NCT04982952
Title: Randomized Trial of a Contingency Management Smoking Cessation Intervention for Homeless Adults
Brief Title: Contingency Management for Smoking Cessation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Tobacco Related Disease Research Program (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 21632; NCI-2021-08359 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2021-07-23; First posted 2021-07-29 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Smoking Cessation; Smoking, Tobacco; Smoking Reduction
Keywords: Contingency Management
MeSH Terms: conditions — Smoking Cessation; Tobacco Smoking; Smoking Reduction

STUDY DESIGN:
Intervention Model Description: Randomization into one of 2 groups will be stratified by recruiter and a binary nicotine dependency code
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Contingency Management (CM) (Experimental): In addition to receiving usual cessation care at the Tom Waddell Urban Health Center (TWUHC), CM intervention participants with CO-verified abstinence will obtain a CM incentive payment, via gift cards and/or cash redeemable in national retail chains.
  Interventions: Behavioral: Contingency Management - Increasing
- Control Group (Other): Participants who choose to attend smoking cessation in the usual care setting at TWUHC will receive a basic $5 payment for attending each study visit.
  Interventions: Behavioral: Fixed payments

INTERVENTIONS:
Behavioral: Contingency Management - Increasing — Increasing incentive payment for abstinent participant
  Arms: Contingency Management (CM)
Behavioral: Fixed payments — Fixed payments for attending study visits
  Arms: Control Group

SUMMARY:
The prevalence of smoking in the homeless population (70%) is over 4 times that of the general population (15%). Homeless adults have not experienced similar declines in tobacco use as the general population has over the past three decades. Homeless adults are interested in smoking cessation and make quit attempts, but are less successful in quitting smoking than the general population. Trials of group behavioral counseling and pharmacotherapy for smoking cessation have not led to substantial long-term abstinence (i.e., abstinence for 6 months or more), suggesting that these interventions alone are insufficient to improve quit rates among homeless adults. Many homeless adults seek health care in safety net clinics; these clinics could bring cessation interventions to scale. Contingency management is a powerful behavior change intervention that reinforces positive health behaviors through the provision of modest incentives (e.g., cash). In this pilot randomized controlled trial, the investigator will test the feasibility and acceptability of a contingency management intervention that provides incentives for smoking cessation for people experiencing homelessness.

DETAILED DESCRIPTION:
In this pilot randomized controlled trial (RCT), the investigator will (1) adapt a known-efficacious extended CM cessation intervention to a novel population and setting, with the ultimate goal of increasing long-term abstinence among homeless adults seeking care in safety net health clinics, (2) develop a corresponding RCT protocol, and (3) conduct a pilot RCT to assess the feasibility and acceptability of the RCT. If the pilot RCT is feasible and acceptable, the investigator will test the adapted intervention in a subsequently-funded, full-scale RCT.

Primary Objectives:

Assess feasibility and acceptability of a CM intervention through:

1. Measuring biochemically-verified point prevalence abstinence at 6 months follow-up.
2. Measuring participant adherence to the protocol.
3. Gathering information on the number of visits attended.
4. Assessing the retention protocol.

Secondary Objectives

Assess feasibility and acceptability of a CM intervention through:

1. Biochemically-verified 7-day point months follow-up at 3 months.
2. Prolonged abstinence at 3 months and 6 months follow-up.
3. Point-prevalent abstinence at 12 months

ELIGIBILITY:
Inclusion Criteria:

1. Are 18 years or older
2. Engaged in care at the Tom Waddell Urban Health Center (TWUHC)
3. Meet criteria for homelessness as defined by the Homeless Emergency Assistance and Rapid Transition to Housing Act
4. Are current smokers (smoked at least 100 cigarettes in lifetime, smoked daily in the past 7 days and at least 5 cigarettes per day, verified by expired Carbon Monoxide (CO) >= 8 parts per million (ppm))
5. Have an intention to quit smoking within the next six months
6. Are attending on-site smoking cessation counseling provided by the behavioral counselors
7. Are English proficient
8. Are able to provide informed consent. Patients who are interested in participating but not enrolled in counseling services will be encouraged to engage in counseling sessions at the time of enrollment.

Exclusion Criteria:

1. Are unable to take nicotine replacement therapy (e.g., pregnancy or myocardial infarction (MI) within the past 2 weeks)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2021-11-09 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Proportion of participants who achieve point prevalence abstinence | 6 months
  The proportion of participants who achieve biochemically-verified 7-day point prevalence abstinence defined as participants (1) reporting not smoking a single cigarette in the past seven days, not even a puff; (2) having carbon monoxide (CO) levels <=5 parts per million (ppm), and (3) urinary anatabine/anabasine assay levels < 2 nanograms per milliliter (ng/ml).
Median number of carbon monoxide (CO) negative samples | 6 months
  The total number of negative CO specimen samples collected throughout the first 6 months of the program will be reported with 24 maximum possible number of samples per person.
Median total number of counseling sessions attended | 6 months
  The number of counseling sessions attended per person will will recorded with a maximum of 5 sessions total.
Proportion of the sample retained as a result of retention procedures over time | Up to 12 months
  The proportion of participants who choose to attend cessation sessions visits at 2 weeks, 1 month, 3 months, 6 months, and 12 months. A participant will be considered lost to follow-up and censored on their last visits if the participants have failed to return for a scheduled visit and the study staff are unable to contact the participant after at least 3 attempts.

SECONDARY OUTCOMES:
Proportion of participants who achieve point prevalence abstinence | 3 months
  The proportion of participants who achieve biochemically-verified 7-day point prevalence abstinence defined as participants (1) reporting not smoking a single cigarette in the past seven days, not even a puff; (2) having carbon monoxide (CO) levels <=5 parts per million (ppm)
Proportion of participants who achieve point prevalence abstinence | 12 months
  The proportion of participants who achieve biochemically-verified 7-day point prevalence abstinence defined as participants (1) reporting not smoking a single cigarette in the past seven days, not even a puff; (2) having carbon monoxide (CO) levels <=5 parts per million (ppm)
Proportion of participants who achieve prolonged abstinence over time | Up to 6 months
  Prolonged abstinence is defined as participants (1) not smoking a single cigarette since the last visit; (2) having CO levels <=5 ppm

CONTACTS AND LOCATIONS:
Overall Officials: Maya Vijayaraghavan, MD, MAS, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - The Richard H. Fine's People's Clinic, San Francisco, California
  - University of California, San Francisco, San Francisco, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Molina MF, Hall SM, Stitzer M, Kushel M, Chakravarty D, Vijayaraghavan M. Contingency management to promote smoking cessation in people experiencing homelessness: Leveraging the electronic health record in a pilot, pragmatic randomized controlled trial. PLoS One. 2022 Dec 16;17(12):e0278870. doi: 10.1371/journal.pone.0278870. eCollection 2022. PMID 36525405